CLINICAL TRIAL: NCT01847300
Title: Computerized Screening and Brief Intervention for Young Military Personnel
Brief Title: cSBI-M for Young Military Personnel
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: bchRFADA13012
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Abuse; Tobacco Dependence; Substance Abuse
Keywords: alcohol abuse; tobacco dependence; substance abuse; SBIRT
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cSBI-M (Experimental): Participants in this group will complete the cSBI-M screening and brief intervention program
  Interventions: Behavioral: cSBI-M
- Treatment as Usual (No Intervention): Participants in this group will receive treatment as usual.

INTERVENTIONS:
Behavioral: cSBI-M — In cSBI-M participants complete a computerized screen for alcohol and tobacco use and then view 10 pages describing the health effects of substance use and true life stories of those affected by substance use.
  Arms: cSBI-M

SUMMARY:
The goal of this project is to test the efficacy of a computer-facilitated Screening and Brief Intervention system adapted for Military use (cSBI-M) in reducing substance use among 18- to 25-yr-old U.S. Navy and U.S. Marine Corps personnel (USN/USMCs). The aims and hypotheses of this project are to: 1)Test the effects of cSBI-M on any alcohol use. Hypothesis: Among 18- to 25-yr-old USN/USMCs coming for routine health screenings, those receiving cSBI-M will have lower rates of any alcohol use at follow-ups compared to TAU. 2) Test the effects of cSBI-M separately as a preventive, early therapeutic, and risk-reduction intervention. Hypotheses: (a) Among 18- to 25-yr-old non-drinking USN/USMCs (negative history of past-12-months drinking at baseline), those receiving cSBI-M will have lower rates of drinking initiation and heavy episodic drinking (HED, a.k.a. "binge" drinking). (b) Among 18- to 25-yr-old drinking USN/USMCs, those receiving cSBI-M will have higher rates of drinking cessation, reduced intensity of drinking (e.g., past-3-months drinking days, HED, and driving after drinking or riding with a drinking driver.(3) Test the effects of cSBI-M on tobacco use; explore its effects on other drug use. (4) Assess potential moderators (e.g., age, gender, race/ethnicity, substance use history +/-, parent/sibling/peer substance use), mediators (e.g., Patient to Provider Connectedness,17 perceived harmfulness of alcohol and drug use), and explore cSBI-M's mechanism of action. Hypotheses: among 12- to 18-yr-old patients coming for routine care, those receiving c-ASBI will have 1) lower rates of any alcohol use, of drinking initiation and riding with a driver who has been drinking, and 2) higher rates of drinking cessation, reduced intensity of drinking, heavy episodic drinking and driving after drinking or riding with a driver who has been drinking.

DETAILED DESCRIPTION:
The goal of this project is to test the efficacy of a computer-facilitated Screening and Brief Intervention system adapted for Military use (cSBI-M) in reducing substance use among 18- to 25-yr-old U.S. Navy and U.S. Marine Corps personnel (USN/USMCs). The aims and hypotheses of this project are to: 1)Test the effects of cSBI-M on any alcohol use. Hypothesis: Among 18- to 25-yr-old USN/USMCs coming for routine health screenings, those receiving cSBI-M will have lower rates of any alcohol use at 3-, 6-, 9- and 12-month follow-ups than Treatment As Usual (TAU). 2) Test the effects of cSBI-M separately as a preventive, early therapeutic, and risk-reduction intervention. Hypotheses: (a) Among 18- to 25-yr-old non-drinking USN/USMCs (negative history of past-12-months drinking at baseline), those receiving cSBI-M will have lower rates of drinking initiation and heavy episodic drinking (HED, a.k.a. "binge" drinking) at 3-, 6-, 9- and 12-month follow-ups than TAU. (b) Among 18- to 25-yr-old drinking USN/USMCs (positive history of past-12-months drinking at baseline), those receiving cSBI-M will have higher rates of drinking cessation, reduced intensity of drinking (e.g., past-3-months drinking days, HED, and driving after drinking or riding with a drinking driver at 3-, 6-, 9- and 12-month follow-ups than TAU. (3) Test the effects of cSBI-M on tobacco use; explore its effects on other drug use. (4) Assess potential moderators (e.g., age, gender, race/ethnicity, substance use history +/-, parent/sibling/peer substance use), mediators (e.g., Patient to Provider Connectedness,17 perceived harmfulness of alcohol and drug use), and explore cSBI-M's mechanism of action. Hypotheses: among 12- to 18-yr-old patients coming for routine care, those receiving c-ASBI will have 1) lower rates of any alcohol use, of drinking initiation and riding with a driver who has been drinking, and 2) higher rates of drinking cessation, reduced intensity of drinking, heavy episodic drinking and driving after drinking or riding with a driver who has been drinking, at 3-, 6-, and 12-month follow-ups compared to Treatment As Usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Navy personnel coming for a routine health screening
* Have email address and internet access for 12-month study period
* Provide informed consent

Exclusion Criteria:

* Unable to read or understand English at a 6th grade level
* Unavailable for 2 of the 4 follow-ups
* Medically or emotionally unstable at the time of the visit

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
alcohol use | past 90 days
  We will measure the past-90-days alcohol use as recorded on the Time-Line-Followback Calendar

SECONDARY OUTCOMES:
Heavy episodic drinking | past-90-days
  We will measure the number of episodes of heavy drinking (binge drinking)
alcohol initiation | past-90-days
  Rates of those initiating drinking in the past 90 days, among those who did not drink at baseline.
Alcohol cessation | Past-90-days
  We will measure the rates of those who stopped drinking in the past-90-days, among those who were drinking at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No